CLINICAL TRIAL: NCT04022070
Title: Short-term Effect of Dynamic Tape ® on Plantar Fascitis; a Pilot Study
Brief Title: The Effect of Dynamic Tape ® on Plantar Fascitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Aurora Castro Mendez, Principal Investigator, University of Seville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 27/02
Record Dates: First submitted 2019-07-05; First posted 2019-07-16 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Fasciitis, Plantar; Foot Tapping
Keywords: foot; fasciitis; tapping
MeSH Terms: conditions — Fasciitis, Plantar; Fasciitis

STUDY DESIGN:
Intervention Model Description: Patients with fasciitis plantar pain
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dynamic Tape (Other): To evaluate the evolution of this symptomatology prior to and thereafter the application of Dynamic Tape® bandage in a sample of subjects affected by plantar fasciitis.
  Interventions: Other: Dynamic Tape® (Tape)

INTERVENTIONS:
Other: Dynamic Tape® (Tape) — To evaluate the evolution of this symptomatology prior to and thereafter the application of Dynamic Tape® bandage affected by plantar fasciitis during a week the Outcome Measure, pain is evaluate with a VAS (visual pain scale).

SUMMARY:
The Dynamic Tape ® (DT) is a new Tape (2009). Dynamic tape ® is a visco-elastic nylon tape material , greater than 200% elastic has manufactured in Asia. The material and adhesive arefast drying and breathable meaning that the tape, if it is correctly applied may stay on for up to 5 days, bearingin mind that if any discomfort, itching, burning, stinging orirritation is felt immediate removal is strongly advised.

Usually tapes are applied in plantar fasciitis to improve the symptoms. The fasciitis plantar is an pain that sometimes incapacitates the physical activity of the patients.

DETAILED DESCRIPTION:
Objective: To evaluate the evolution of this symptomatology prior to and thereafter the application of Dynamic Tape® bandage in a sample of 15 amateur athletes affected by plantar fasciitis. The assessment will be performed using an analogue visual scale (EVA). Material and methods: the aim of the study is to evaluate a group of 15 amateur athletic subjects , all individuals suffering plantar fasciitis without any previous or current treatment. The age, from 18 to 65 years old. Samplings will be performed intentionally without a control group.

The control group will use a Low-dye tape and will be evaluated before and after a week

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of fasciitis
* Plantar fasciitis pain

Exclusion Criteria:

Current treatment of fasciitis pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Plantar fasciitis pain | 7 days
  Evaluation before and after a week of use of a Dynamic Tape. Visual analogic scale.
  The visual analogue scale (VAS) is commonly used as the outcome measure for such studies. It is usually presented as a 100-mm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "no pain at all" and "worst pain imaginable." The Primary and second Outcome Measures (pain, VAS) . Time Frame includes more than one time point. The initial evaluation, the day of inclusion in the study and the second one a week after the use of the tape

CONTACTS AND LOCATIONS:
Locations (1):
- Aurora Castro Mendez, Seville, Spain

IPD SHARING:
Plan to Share IPD: Undecided